CLINICAL TRIAL: NCT00978120
Title: A Phase II Study in Patients With Asthma to Assess the Safety and Immunogenicity of an Unadjuvanted Novartis H1N1 Influenza Vaccine Administered at Two Dose Levels
Brief Title: Safety and Efficacy of an H1N1 Influenza Vaccine in People With Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: DAIT-AAIB-flu-001
Record Dates: First submitted 2009-09-15; First posted 2009-09-16 (Estimated); Results first posted 2012-08-06 (Estimated); Last update posted 2012-08-10 (Estimated); Status verified 2012-08

CONDITIONS: H1N1 Influenza Virus
Keywords: Influenza A Virus, H1N1 Subtype; Vaccine

ARMS (2):
- H1N1 vaccine high dose (Experimental): Participants will be stratified according to asthma severity and will receive the high dosage of the H1N1 vaccine.
  Interventions: Biological: H1N1 vaccine high dose
- H1N1 vaccine low dose (Experimental): Participants will be stratified according to asthma severity and will receive the low dosage of the H1N1 vaccine.
  Interventions: Biological: H1N1 vaccine low dose

INTERVENTIONS:
Biological: H1N1 vaccine high dose — 30 mcg of unadjuvanted Novartis H1N1 vaccine delivered as two, 15 micrograms (mcg), intramuscular injections. Each 30 mcg dose is administered 21 days apart.
  Arms: H1N1 vaccine high dose
Biological: H1N1 vaccine low dose — 15 mcg of unadjuvanted Novartis H1N1 vaccine delivered in two intramuscular injections 21 days apart
  Arms: H1N1 vaccine low dose

SUMMARY:
The purpose of this study is to assess the safety and the body's immune response (body's defense against disease) to an experimental H1N1 influenza vaccine in people with asthma. The study will enroll 350, and possibly up to 400 healthy adults ages 12 and older with mild, moderate, or severe asthma. Participants will be randomly assigned to 1 of 2 possible vaccine groups: group 1 will receive 15 mcg of H1N1 vaccine; group 2 will receive 30 mcg of H1N1 vaccine given as two 15 mcg injections. Both groups will receive vaccine injections on days 0 and 21.

Study procedures include: medical history, physical exam, spirometry, maintaining a memory aid and, and blood sample collection. Participants will be involved in study related procedures for approximately 7 months.

DETAILED DESCRIPTION:
A new swine-origin influenza A/H1N1 virus was recently identified as a significant cause of respiratory illness in Mexico and the United States. In response, the World Health Organization (WHO) declared a pandemic on June 11, 2009. Current data indicates that licensed seasonal influenza vaccines are not likely to provide protection against the new H1N1 virus. Development and deployment of a vaccine for the new H1N1 virus, particularly to at-risk populations, is essential.

Groups at risk for influenza yearly include the elderly and those with asthma, and current guidelines from the Advisory Committee on Immunization Practices (ACIP) recommend vaccination of adults and children with asthma. Early, unpublished data on US patients hospitalized by H1N1 infection indicates that many had underlying asthma, and it is expected people with asthma will be on a priority list for H1N1 influenza vaccination. Data also indicate that increased dosage of vaccines may increase development of antibodies and that use of certain inhalers may affect immunization. This study will test the safety and immunogenicity of an unadjuvanted, inactivated H1N1 vaccine at two dosage levels in people with asthma.

Participation in this study will last approximately 34 weeks. Participants will be stratified into two groups: those with mild to moderate versus those with severe asthma. All participants will be randomly assigned to receive either a high dose (30 mcg) or low dose (15 mcg) H1N1 vaccine. Both vaccine dosages will be administered in two intramuscular injections 21 days apart. Participants assigned to the higher dose (30 mcg) will receive two injections of the 15 mcg vaccine at each administration.

Participants will complete study visits at entry, administration of the vaccines on Days 1 and 21, follow-ups a week after each vaccine injection, and 21 days after the second injection. Measurements at these visits will include spirometry (measurement of air entering and leaving the lungs), a questionnaire about asthma, a targeted physical examination, an adverse event and medication assessment, inspection of vaccination site, and collection of a blood sample. A urine sample will be collected for pregnancy test before each vaccination. In additions, for 8 days after each vaccination injection participants will keep a diary recording oral temperature, adverse events, asthma symptoms, and use of inhalers. These diaries will be reviewed at study visits. Participants will also receive follow-up phone calls to assess safety 60, 120, and 180 days after the last vaccine injection.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of mild/moderate or severe asthma according to Severe Asthma Research Project (SARP) definitions and either a SARP participant or having prior participation in the studies or clinics of the investigators
* Males and females age 12 (inclusive) and older
* Females of child-bearing potential must not be pregnant and must agree to practice adequate contraception that may include, but is not limited to: abstinence, monogamous relationship with vasectomized partner, barrier methods such as condoms, diaphragms, spermicides, intrauterine devices, and licensed hormonal methods during the study for at least 30 days following the last vaccination.
* Able to understand and comply with planned study procedures
* Will provide written informed consent and assent (if age appropriate) prior to initiation of any study procedures

Exclusion Criteria:

* Allergy to eggs or other components of the vaccine, including gelatin, formaldehyde, octoxinol, thimerosal, and chicken protein
* Positive urine pregnancy test within 24 hours prior to vaccination, if a female of childbearing potential
* Currently breastfeeding
* History of smoking 20 pack-years or greater (current or former smokers with a history of less than 20 pack-years can be included in the study)
* Has been previously diagnosed by a physician with chronic obstructive pulmonary disease, chronic bronchitis, emphysema, or cystic fibrosis
* Has received anticancer chemotherapy or radiation therapy (cytotoxic) within the past 36 months
* Has an active neoplastic disease or a history of any hematologic malignancy
* Has a diagnosis of schizophrenia, bipolar disease, or other major psychiatric diagnosis
* Has been hospitalized for psychiatric illness, history of suicide attempt, or confinement for danger to self or others within the past 10 years
* Receiving psychiatric drugs (subjects who are receiving a single antidepressant drug and are stable for at least 3 months prior to study entry, without de-compensating symptoms, will be allowed to enroll)
* History of receiving immunoglobulin, including anti-cytokine antibodies, or other blood product within the 3 months prior to vaccination in this study
* Has received an experimental agent (vaccine, drug, biologic, device, blood product, or medication) within 1 month prior to vaccination in this study or expect to receive an experimental agent during this study (prior to the Day 141 follow-up call - 100 days after the second vaccination)
* Has received any live licensed vaccines within 4 weeks or inactivated licensed vaccines within 2 weeks prior to vaccination in this study, or plan receipt of such vaccines within 21 days following the second vaccination
* Has a history of severe reactions following previous immunization with influenza virus vaccines
* Has an acute illness, including an oral temperature greater than 100.4°F, within 1 week of either vaccination
* Has a chronic neurologic or autoimmune disorder
* Has a history of Guillain-Barré Syndrome
* Has an acute or chronic medical condition that, in the opinion of the investigator, would render vaccination unsafe, or would interfere with the evaluation of vaccine response
* Has an ongoing asthma exacerbation or had an asthma exacerbation that was resolved less than 7 days prior to vaccination
* Has any condition that would, in the opinion of the site investigator, place the participant at an unacceptable risk of injury, render the participant unable to meet the requirements of the protocol, or interfere with the successful completion of the study.
* Participated in a novel influenza H1N1 2009 vaccine study in the past two years or has a history of novel influenza H1N1 2009 infection or treatment
* Has known active HIV, Hepatitis B or Hepatitis C infection
* Has a history of alcohol or drug abuse in the last 5 years
* Plans to travel outside of North America in the time between the first vaccination and 42 days following the first vaccination
* Does not speak English primarily

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 390 (Actual)
Dates: Start 2009-10; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Busse, MD, Principal Investigator — University of Wisconsin Medical School
Locations (7):
- United States (7):
  - Emory University, Atlanta, Georgia
  - Washington University School of Medicine, St Louis, Missouri
  - Wake Forest University School of Medicine, Winston-Salem, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - University of Pittsburgh Asthma Institute, Pittsburgh, Pennsylvania
  - University of Virginia, Charlottesville, Virginia
  - University of Wisconsin, Madison, Wisconsin

REFERENCES:
- [Background] Novel Swine-Origin Influenza A (H1N1) Virus Investigation Team; Dawood FS, Jain S, Finelli L, Shaw MW, Lindstrom S, Garten RJ, Gubareva LV, Xu X, Bridges CB, Uyeki TM. Emergence of a novel swine-origin influenza A (H1N1) virus in humans. N Engl J Med. 2009 Jun 18;360(25):2605-15. doi: 10.1056/NEJMoa0903810. Epub 2009 May 7. PMID 19423869
- [Background] Patriarca PA, Cox NJ. Influenza pandemic preparedness plan for the United States. J Infect Dis. 1997 Aug;176 Suppl 1:S4-7. doi: 10.1086/514174. PMID 9240686
- [Background] Proceedings of the ATS workshop on refractory asthma: current understanding, recommendations, and unanswered questions. American Thoracic Society. Am J Respir Crit Care Med. 2000 Dec;162(6):2341-51. doi: 10.1164/ajrccm.162.6.ats9-00. No abstract available. PMID 11112161
- [Result] Busse WW, Peters SP, Fenton MJ, Mitchell H, Bleecker ER, Castro M, Wenzel S, Erzurum SC, Fitzpatrick AM, Teague WG, Jarjour N, Moore WC, Sumino K, Simeone S, Ratanamaneechat S, Penugonda M, Gaston B, Ross TM, Sigelman S, Schiepan JR, Zaccaro DJ, Crevar CJ, Carter DM, Togias A. Vaccination of patients with mild and severe asthma with a 2009 pandemic H1N1 influenza virus vaccine. J Allergy Clin Immunol. 2011 Jan;127(1):130-7, 137.e1-3. doi: 10.1016/j.jaci.2010.11.014. Epub 2010 Dec 9. PMID 21145578

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants were recruited from October 16 to November 13, 2009 at the seven National Heart, Lung, and Blood Institute (NHLBI)- funded Severe Asthma Research Program sites.
Groups:
- Mild/Moderate Asthma, Low Dose Vaccine (15mcg): Participants with mild-to-moderate asthma received one 15 micrograms (mcg) dose of unadjuvanted,[1] inactivated Novartis H1N1 pandemic influenza vaccine by intramuscular injection on Day 1 and Day 21.
- Mild/Moderate Asthma, High Dose Vaccine (30mcg): Participants with mild-to-moderate asthma received two 15 mcg doses of unadjuvanted,[1] inactivated Novartis H1N1 pandemic influenza vaccine by intramuscular injections on Day 1 and Day 21.
- Severe Asthma, Low Dose Vaccine (15mcg): Participants with severe asthma received one 15 mcg dose of unadjuvanted,[1] inactivated Novartis H1N1 pandemic influenza vaccine by intramuscular injection on Day 1 and Day 21.
- Severe Asthma, High Dose Vaccine (30mcg): Participants with severe asthma received two 15 mcg doses of unadjuvanted,[1] inactivated Novartis H1N1 pandemic influenza vaccine by intramuscular injections on Day 1 and Day 21.
  [1] Unadjuvanted: No agents added to, or used in conjunction with, vaccine antigens to augment or potentiate (and possibly target) the specific immune response to the antigen. (U.S. Food And Drug Administration)
Period: Overall Study
Arm/Group | Mild/Moderate Asthma, Low Dose Vaccine (15mcg) | Mild/Moderate Asthma, High Dose Vaccine (30mcg) | Severe Asthma, Low Dose Vaccine (15mcg) | Severe Asthma, High Dose Vaccine (30mcg)
Started | 110 | 107 | 87 | 86
Completed | 108 | 107 | 84 | 84
Not Completed | 2 | 0 | 3 | 2
Not completed — Death | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 3 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0 | 0
Not completed — Moved out of state | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mild/Moderate Asthma, Low Dose Vaccine (15mcg) | Mild/Moderate Asthma, High Dose Vaccine (30mcg) | Severe Asthma, Low Dose Vaccine (15mcg) | Severe Asthma, High Dose Vaccine (30mcg) | Total
Number analyzed (Participants) | 110 | 107 | 87 | 86 | 390
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 22 | 23 | 12 | 10 | 67
  Between 18 and 65 years | 80 | 79 | 67 | 68 | 294
  >=65 years | 8 | 5 | 8 | 8 | 29
Age Continuous [Mean (Standard Deviation); unit: years] | 39.1 (18.1) | 36.3 (17.0) | 45.2 (17.0) | 46.5 (17.3) | 41.3 (17.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 72 | 62 | 52 | 45 | 231
  Male | 38 | 45 | 35 | 41 | 159
Region of Enrollment [Number; unit: participants]
  United States | 110 | 107 | 87 | 86 | 390
Age at Asthma Onset [Mean (Standard Deviation); unit: years] — The age at asthma onset is the age defined in years when the participant was told by a physician that he/she has asthma. This was calculated by subtracting the participant's age at the baseline visit (visit 1) from the number of years the participant reported to have known having asthma.
  years | 17.1 (17.0) | 16.4 (14.9) | 21.9 (19.7) | 21.9 (20.1) | 19.0 (17.9)
Asthma Duration [Mean (Standard Deviation); unit: years] — Asthma duration is the number of years since the participant was told by a physician that he/she has asthma as reported at the baseline visit, visit 1.
  years | 21.9 (13.9) | 19.9 (13.4) | 23.3 (16.5) | 24.6 (17.8) | 22.3 (15.3)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — BMI is a number calculated from a person's height and weight that provides a reliable indicator of body fatness for most people. Higher values reflect greater amount of body fat. [1] In adults, a BMI less than 18.5 is underweight; 18.5 to 24.9 is a normal or healthy weight; greater than or equal to 25.0 is overweight. The height and weight was collected at baseline only.
  [1]: Healthy Weight , Assessing Your Weight , Body Mass Index http://www.cdc.gov/healthyweight/assessing/bmi/index.html
  kg/m^2 | 29.5 (8.5) | 28.5 (6.8) | 31.8 (9.7) | 30.1 (8.0) | 29.9 (8.3)
Forced Expiratory Volume in 1 second (FEV1) % Predicted [Mean (Standard Deviation); unit: percentage] — FEV1 is air volume exhaled in 1 second during spirometry. Asthma severity classification for trial: mild--pre-bronchodilator FEV1 ≥ 80% predicted requiring no/ low-moderate dose of inhaled glucocorticoids; moderate--pre-bronchodilator FEV1 <80% predicted requiring no/ low-moderate dose of inhaled glucocorticoids; severe--requiring high-dose inhaled glucocorticoids with/without continuous/near continuous oral glucocorticoids, or uncontrolled despite treatment. FEV1 percent of predicted value is FEV1 converted to a percentage of normal, based on height, weight, and race.
  percentage | 83.8 (16.3) | 86.6 (17.6) | 72.6 (19.4) | 69.8 (20.8) | 79.0 (19.7)
Forced Vital Capacity (FVC) % Predicted [Mean (Standard Deviation); unit: percentage] — FVC is a lung function test that measures the total amount of air exhaled. The percent of predicted value is FVC converted to a percentage of normal, based on height, weight, and race. Estimates of severity of abnormalities in flow volume measured by FVC: Mild-65-80% of predicted value; Moderate-50-65% of predicted value; Severe-<50% of predicted value.
  percentage | 92.6 (14.3) | 94.3 (16.1) | 85.0 (17.1) | 80.9 (18.7) | 88.8 (17.3)
FEV1/FVC Ratio [Mean (Standard Deviation); unit: Ratio (x 100)] — The FEV1 (forced expiratory volume 1))/ FVC (forced vital capacity) ratio is used to evaluate airways obstructions since pure restrictive ventilatory defects cause an equal reduction in the FEV1 and the FVC. An FEV1/FVC ratio below 80% indicates airflow obstruction. Normal FEV1/FVC: 8 - 19 years of age=85%; 20-39 years of age=80%; 40- 59 years of age 75%; 60-80 years of age 70% [1]
  [1]: National Asthma Education and Prevention Program Expert Panel Report 3, Guidelines for the Diagnosis and Management of Asthma. Oct. 2007. http://www.nhlbi.nih.gov/guidelines/asthma/asthsumm.pdf
  Ratio (x 100) | 74.5 (9.07) | 75.7 (8.99) | 68.4 (10.91) | 68.4 (11.76) | 72.1 (10.62)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Serious Adverse Events (SAEs) Attributed To Vaccination
Description: Percentage of participants with serious adverse events (SAEs) attributed to vaccination, as determined by site investigators at the time of reporting.
Time Frame: Measured at Baseline Visit and Days 1, 8, 21, 28, 41, 80, 120, and 201
Measure: Number; unit: percentage of participants
Arm/Group | Mild/Moderate Asthma, Low Dose Vaccine (15mcg) | Mild/Moderate Asthma, High Dose Vaccine (30mcg) | Severe Asthma, Low Dose Vaccine (15mcg) | Severe Asthma, High Dose Vaccine (30mcg)
Number analyzed (Participants) | 110 | 107 | 87 | 86
percentage of participants | 1 | 0 | 3 | 0

2. Primary Outcome: Percentage of Participants With Reactogenicity Adverse Events (AEs) Status Post Vaccine 1
Description: Percentage of participants with reactogenicity AEs, local (erythema, ecchymosis, induration, pain and tenderness at the injection sites) and systemic (feverishness, chills, fatigue, myalgias, arthralgias, headache and nausea), within 8 Days After Vaccination 1 by Dose Level Group.
Time Frame: Days 1 through 8
Measure: Number; unit: percentage of participants
Arm/Group | Mild/Moderate Asthma, Low Dose Vaccine (15mcg) | Mild/Moderate Asthma, High Dose Vaccine (30mcg) | Severe Asthma, Low Dose Vaccine (15mcg) | Severe Asthma, High Dose Vaccine (30mcg)
Number analyzed (Participants) | 110 | 107 | 87 | 86
percentage of participants
  Systemic | 58 | 63 | 64 | 74
  Local | 55 | 54 | 33 | 52
Statistical Analysis 1: Comparison: Mild/Moderate Asthma, Low Dose Vaccine (15mcg) vs Mild/Moderate Asthma, High Dose Vaccine (30mcg) vs Severe Asthma, Low Dose Vaccine (15mcg) vs Severe Asthma, High Dose Vaccine (30mcg); Test type: Superiority or Other; p = 0.014, Fisher Exact

3. Primary Outcome: Percentage of Participants With Reactogenicity Adverse Events (AEs) Status Post Vaccine 2
Description: Percentage of participants with reactogenicity AEs, local (erythema, ecchymosis, induration, pain and tenderness at the injection sites) and systemic (feverishness, chills, fatigue, myalgias, arthralgias, headache and nausea), within 8 Days After Vaccination 2 by Dose Level Group.
Time Frame: Days 21 through 28
Measure: Number; unit: percentage of participants
Arm/Group | Mild/Moderate Asthma, Low Dose Vaccine (15mcg) | Mild/Moderate Asthma, High Dose Vaccine (30mcg) | Severe Asthma, Low Dose Vaccine (15mcg) | Severe Asthma, High Dose Vaccine (30mcg)
Number analyzed (Participants) | 102 | 99 | 80 | 76
percentage of participants
  Systemic | 47 | 47 | 48 | 42
  Local | 46 | 60 | 29 | 38
Statistical Analysis 1: Comparison: Mild/Moderate Asthma, Low Dose Vaccine (15mcg) vs Mild/Moderate Asthma, High Dose Vaccine (30mcg) vs Severe Asthma, Low Dose Vaccine (15mcg) vs Severe Asthma, High Dose Vaccine (30mcg); Test type: Superiority or Other; p = 0.05, Fisher Exact

4. Primary Outcome: Percentage of Participants With Asthma Exacerbations Status Post Vaccine 1
Description: Percentage of participants with asthma exacerbations within 8 days after vaccination 1. Any of the following events are considered asthma exacerbation: Increase in the daily use of bronchodilator rescue medication for 2 consecutive days; an increase is defined as ≥6puffs of bronchodilator from a metered-dose inhaler or ≥2 uses of nebulized albuterol above average use reported in the two weeks prior to Visit 1. Increase in use of systemic corticosteroids or the addition of systemic corticosteroids to treatment regimen for asthma. Unscheduled use of health care for the treatment of asthma.
Time Frame: Days 1 to 8
Measure: Number; unit: percentage of participants
Arm/Group | Mild/Moderate Asthma, Low Dose Vaccine (15mcg) | Mild/Moderate Asthma, High Dose Vaccine (30mcg) | Severe Asthma, Low Dose Vaccine (15mcg) | Severe Asthma, High Dose Vaccine (30mcg)
Number analyzed (Participants) | 110 | 107 | 87 | 86
percentage of participants | 4 | 2 | 8 | 3

5. Primary Outcome: Percentage of Participants With Asthma Exacerbations Status Post Vaccination 2
Description: Percentage of participants with asthma exacerbations within 8 days after vaccination 2. Any of the following events are considered asthma exacerbation: Increase in the daily use of bronchodilator rescue medication for 2 consecutive days; an increase is defined as ≥6puffs of bronchodilator from a metered-dose inhaler or ≥2 uses of nebulized albuterol above average use reported in the two weeks prior to Visit 1. Increase in use of systemic corticosteroids or the addition of systemic corticosteroids to treatment regimen for asthma. Unscheduled use of health care for the treatment of asthma.
Time Frame: Days 21 to 28
Measure: Number; unit: percentage of participants
Arm/Group | Mild/Moderate Asthma, Low Dose Vaccine (15mcg) | Mild/Moderate Asthma, High Dose Vaccine (30mcg) | Severe Asthma, Low Dose Vaccine (15mcg) | Severe Asthma, High Dose Vaccine (30mcg)
Number analyzed (Participants) | 102 | 99 | 80 | 76
percentage of participants | 4 | 1 | 3 | 6

6. Secondary Outcome: Percentage of Participants With Seroconversion at Day 21 Following Single Administration of Vaccination, Mild-Moderate Asthmatics
Description: Percentage of participants with seroconversion defined as a four-fold or greater hemagglutination inhibition assay (HAI) antibody titer increase compared to baseline against the novel influenza hemagglutinin type 1 and neuraminidase type 1 (H1N1) 2009 virus following a single administration of Novartis H1N1 vaccine at each dose, combined across age groups.
Time Frame: Days 1 to 21
Measure: Number; unit: percentage of participants
Groups:
- Mild/Moderate Asthma, Low Dose Vaccine (15mcg): Participants with mild-to-moderate asthma received one 15 micrograms (mcg) dose of unadjuvanted[1], inactivated Novartis H1N1 pandemic influenza vaccine by intramuscular injection on Day 1 and Day 21.
- Mild/Moderate Asthma, High Dose Vaccine (30mcg): Participants with mild-to-moderate asthma received two 15 mcg doses of unadjuvanted[1], inactivated Novartis H1N1 pandemic influenza vaccine by intramuscular injections on Day 1 and Day 21.
  [1] Unadjuvanted: No agents added to, or used in conjunction with, vaccine antigens to augment or potentiate (and possibly target) the specific immune response to the antigen. (U.S. Food And Drug Administration)
Arm/Group | Mild/Moderate Asthma, Low Dose Vaccine (15mcg) | Mild/Moderate Asthma, High Dose Vaccine (30mcg)
Number analyzed (Participants) | 107 | 107
percentage of participants | 80.4 | 85.0
Statistical Analysis 1: Comparison: Mild/Moderate Asthma, Low Dose Vaccine (15mcg) vs Mild/Moderate Asthma, High Dose Vaccine (30mcg); Test type: Superiority or Other; p = 0.470, Fisher Exact

7. Secondary Outcome: Percentage of Participants With Seroconversion at Day 21 Following Single Administration of Vaccination, Severe Asthmatics
Description: Percentage of participants with seroconversion defined as a four-fold or greater hemagglutination inhibition assay(HAI) antibody titer increase compared to baseline against the novel influenza hemagglutinin type 1 and neuraminidase type 1 (H1N1) 2009 virus following a single administration of Novartis H1N1 vaccine at each dose, combined across age groups.
Time Frame: Days 1 to 21
Measure: Number; unit: percentage of participants
Groups:
- Severe Asthma, Low Dose Vaccine (15mcg): Participants with severe asthma received one 15 mcg dose of unadjuvanted[1], inactivated Novartis H1N1 pandemic influenza vaccine by intramuscular injection on Day 1 and Day 21.
- Severe Asthma, High Dose Vaccine (30mcg): Participants with severe asthma received two 15 mcg doses of unadjuvanted[1], inactivated Novartis H1N1 pandemic influenza vaccine by intramuscular injections on Day 1 and Day 21.
  [1] Unadjuvanted: No agents added to, or used in conjunction with, vaccine antigens to augment or potentiate (and possibly target) the specific immune response to the antigen. (U.S. Food And Drug Administration)
Arm/Group | Severe Asthma, Low Dose Vaccine (15mcg) | Severe Asthma, High Dose Vaccine (30mcg)
Number analyzed (Participants) | 86 | 85
percentage of participants | 75.6 | 85.9
Statistical Analysis 1: Comparison: Severe Asthma, Low Dose Vaccine (15mcg) vs Severe Asthma, High Dose Vaccine (30mcg); Test type: Superiority or Other; p = 0.120, Fisher Exact

8. Secondary Outcome: Percentage of Participants With Seroprotection at Day 21 Following Single Administration of Vaccination, Mild-Moderate Asthmatics
Description: Percentage of participants with seroprotection defined as hemagglutination inhibition assay (HAI) antibody titer of 1:40 or greater against influenza H1N1 2009 virus following a single administration of the H1N1 vaccine at each dose, combined across age groups.
Time Frame: Days 1 to 21
Measure: Number; unit: percentage of participants
Arm/Group | Mild/Moderate Asthma, Low Dose Vaccine (15mcg) | Mild/Moderate Asthma, High Dose Vaccine (30mcg)
Number analyzed (Participants) | 107 | 107
percentage of participants | 90.7 | 95.3
Statistical Analysis 1: Comparison: Mild/Moderate Asthma, Low Dose Vaccine (15mcg) vs Mild/Moderate Asthma, High Dose Vaccine (30mcg); Test type: Superiority or Other; p = 0.284, Fisher Exact

9. Secondary Outcome: Percentage of Participants With Seroprotection at Day 21 Following Single Administration of Vaccination, Severe Asthmatics
Description: as for outcome 8
Time Frame: Days 1 to 21
Measure: Number; unit: percentage of participants
Arm/Group | Severe Asthma, Low Dose Vaccine (15mcg) | Severe Asthma, High Dose Vaccine (30mcg)
Number analyzed (Participants) | 86 | 85
percentage of participants | 77.9 | 94.1
Statistical Analysis 1: Comparison: Severe Asthma, Low Dose Vaccine (15mcg) vs Severe Asthma, High Dose Vaccine (30mcg); Test type: Superiority or Other; p = 0.004, Fisher Exact

10. Primary Outcome: Percentage of Participants With Seroconversion at Day 28 Following Two Administrations of Vaccination, Mild-Moderate Asthmatics
Description: Seroconversion: The percentage of participants with a four-fold or greater hemagglutination inhibition assay (HAI) antibody titer increase compared to baseline against the novel influenza hemagglutinin type 1 and neuraminidase type 1 (H1N1) 2009 virus following two administrations of Novartis H1N1 vaccine at each dose, combined across age groups.
Time Frame: Days 1 to 28
Measure: Number; unit: percentage of participants
Arm/Group | Mild/Moderate Asthma, Low Dose Vaccine (15mcg) | Mild/Moderate Asthma, High Dose Vaccine (30mcg)
Number analyzed (Participants) | 103 | 97
percentage of participants | 80.6 | 86.6
Statistical Analysis 1: Comparison: Mild/Moderate Asthma, Low Dose Vaccine (15mcg) vs Mild/Moderate Asthma, High Dose Vaccine (30mcg); Test type: Superiority or Other; p = 0.341, Fisher Exact

11. Primary Outcome: Percentage of Participants With Seroconversion at Day 28 Following Two Administrations of Vaccination, Severe Asthmatics
Description: as for outcome 10
Time Frame: Days 1 to 28
Measure: Number; unit: percentage of participants
Arm/Group | Severe Asthma, Low Dose Vaccine (15mcg) | Severe Asthma, High Dose Vaccine (30mcg)
Number analyzed (Participants) | 77 | 76
percentage of participants | 68.8 | 85.5
Statistical Analysis 1: Comparison: Severe Asthma, Low Dose Vaccine (15mcg) vs Severe Asthma, High Dose Vaccine (30mcg); Test type: Superiority or Other; p = 0.020, Fisher Exact

12. Primary Outcome: Percentage of Participants With Seroconversion at Day 41 Following Two Administrations of Vaccination, Mild-Moderate Asthmatics
Description: as for outcome 10
Time Frame: Days 1 to 41
Measure: Number; unit: percentage of participants
Arm/Group | Mild/Moderate Asthma, Low Dose Vaccine (15mcg) | Mild/Moderate Asthma, High Dose Vaccine (30mcg)
Number analyzed (Participants) | 103 | 99
percentage of participants | 73.8 | 80.8
Statistical Analysis 1: Comparison: Mild/Moderate Asthma, Low Dose Vaccine (15mcg) vs Mild/Moderate Asthma, High Dose Vaccine (30mcg); Test type: Superiority or Other; p = 0.245, Fisher Exact

13. Primary Outcome: Percentage of Participants With Seroconversion at Day 41 Following Two Administrations of Vaccination, Severe Asthmatics
Description: as for outcome 10
Time Frame: Days 1 to 41
Measure: Number; unit: percentage of participants
Arm/Group | Severe Asthma, Low Dose Vaccine (15mcg) | Severe Asthma, High Dose Vaccine (30mcg)
Number analyzed (Participants) | 76 | 76
percentage of participants | 72.4 | 82.9
Statistical Analysis 1: Comparison: Severe Asthma, Low Dose Vaccine (15mcg) vs Severe Asthma, High Dose Vaccine (30mcg); Test type: Superiority or Other; p = 0.173, Fisher Exact

14. Primary Outcome: Percentage of Participants With Seroprotection at Day 28 Following Two Administrations of Vaccination, Mild-Moderate Asthmatics
Description: Seroprotection: The percentage of participants with a hemagglutination inhibition assay (HAI) antibody titer of 1:40 or greater against influenza H1N1 2009 virus following two administrations of the H1N1 vaccine at each dose, combined across age groups.
Time Frame: Days 1 to 28
Measure: Number; unit: percentage of participants
Arm/Group | Mild/Moderate Asthma, Low Dose Vaccine (15mcg) | Mild/Moderate Asthma, High Dose Vaccine (30mcg)
Number analyzed (Participants) | 103 | 97
percentage of participants | 87.4 | 91.8
Statistical Analysis 1: Comparison: Mild/Moderate Asthma, Low Dose Vaccine (15mcg); Test type: Superiority or Other; p = 0.362, Fisher Exact

15. Primary Outcome: Percentage of Participants With Seroprotection at Day 28 Following Two Administrations of Vaccination, Severe Asthmatics
Description: Percentage of participants with seroprotection defined as a hemagglutination inhibition assay (HAI) antibody titer of 1:40 or greater against influenza H1N1 2009 virus following two administrations of the H1N1 vaccine at each dose, combined across age groups.
Time Frame: Days 1 to 28
Measure: Number; unit: percentage of participants
Arm/Group | Severe Asthma, Low Dose Vaccine (15mcg) | Severe Asthma, High Dose Vaccine (30mcg)
Number analyzed (Participants) | 77 | 76
percentage of participants | 76.6 | 93.4
Statistical Analysis 1: Comparison: Severe Asthma, Low Dose Vaccine (15mcg) vs Severe Asthma, High Dose Vaccine (30mcg); Test type: Superiority or Other; p = 0.006, Fisher Exact

16. Primary Outcome: Percentage of Participants With Seroprotection at Day 41 Following Two Administrations of Vaccination, Mild-Moderate Asthmatics
Description: as for outcome 15
Time Frame: Days 1 to 41
Measure: Number; unit: percentage of participants
Arm/Group | Mild/Moderate Asthma, Low Dose Vaccine (15mcg) | Mild/Moderate Asthma, High Dose Vaccine (30mcg)
Number analyzed (Participants) | 103 | 99
percentage of participants | 82.5 | 93.9
Statistical Analysis 1: Comparison: Mild/Moderate Asthma, Low Dose Vaccine (15mcg) vs Mild/Moderate Asthma, High Dose Vaccine (30mcg); Test type: Superiority or Other; p = 0.016, Fisher Exact

17. Primary Outcome: Percentage of Participants With Seroprotection at Day 41 Following Two Administrations of Vaccination, Severe Asthmatics
Description: as for outcome 15
Time Frame: Days 1 to 41
Measure: Number; unit: percentage of participants
Arm/Group | Severe Asthma, Low Dose Vaccine (15mcg) | Severe Asthma, High Dose Vaccine (30mcg)
Number analyzed (Participants) | 76 | 76
percentage of participants | 75.0 | 89.5
Statistical Analysis 1: Comparison: Severe Asthma, Low Dose Vaccine (15mcg) vs Severe Asthma, High Dose Vaccine (30mcg); Test type: Superiority or Other; p = 0.032, Fisher Exact

ADVERSE EVENTS:
Time Frame: Enrollment through last day of followup (Day 201, target last day)
Groups:
- Mild/Moderate Asthma, Low Dose Vaccine (15 Mcg): Participants with mild/moderate asthma received one 15 mcg dose of unadjuvanted, inactivated Novartis H1N1 pandemic influenza vaccine by intramuscular injection on Day 1 and Day 21.
- Mild/Moderate Asthma, High Dose Vaccine (30mcg): Participants with mild/moderate asthma received two 15 mcg doses of unadjuvanted, inactivated Novartis H1N1 pandemic influenza vaccine by intramuscular injection on Day 1 and Day 21.
- Severe Asthma, Low Dose Vaccine (15mcg): Participants with severe asthma received one 15 mcg dose of unadjuvanted, inactivated Novartis H1N1 pandemic influenza vaccine by intramuscular injection on Day 1 and Day 21.
- Severe Asthma, High Dose Vaccine (30mcg): Participants with severe asthma received two 15 mcg doses of unadjuvanted, inactivated Novartis H1N1 pandemic influenza vaccine by intramuscular injection on Day 1 and Day 21.
Arm/Group | Mild/Moderate Asthma, Low Dose Vaccine (15 Mcg) | Mild/Moderate Asthma, High Dose Vaccine (30mcg) | Severe Asthma, Low Dose Vaccine (15mcg) | Severe Asthma, High Dose Vaccine (30mcg)
Serious Adverse Events (participants affected / at risk) | 4/110 | 4/107 | 12/87 | 6/86
Other Adverse Events (participants affected / at risk) | 29/110 | 15/107 | 25/87 | 25/86
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mild/Moderate Asthma, Low Dose Vaccine (15 Mcg) (N=110) | Mild/Moderate Asthma, High Dose Vaccine (30mcg) (N=107) | Severe Asthma, Low Dose Vaccine (15mcg) (N=87) | Severe Asthma, High Dose Vaccine (30mcg) (N=86)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abasia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Localised infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 7 (7) | 3 (3)
Drug rehabilitation (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hysterectomy (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mild/Moderate Asthma, Low Dose Vaccine (15 Mcg) (N=110) | Mild/Moderate Asthma, High Dose Vaccine (30mcg) (N=107) | Severe Asthma, Low Dose Vaccine (15mcg) (N=87) | Severe Asthma, High Dose Vaccine (30mcg) (N=86)
Upper respiratory tract infection (Infections and infestations) | 12 (12) | 9 (9) | 11 (11) | 8 (8)
Forced expiratory volume decreased (Investigations) | 4 (4) | 1 (2) | 7 (9) | 8 (13)
Asthma (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 3 (4) | 10 (11) | 9 (9)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 4 (4) | 1 (1) | 5 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No